CLINICAL TRIAL: NCT02207634
Title: A Double-Blind, Placebo Controlled, Multicenter Study to Assess the Effect of Evolocumab on Cognitive Function in Patients With Clinically Evident Cardiovascular Disease and Receiving Statin Background Lipid Lowering Therapy: A Study for Subjects Enrolled in the FOURIER (Study 20110118) Trial
Brief Title: Evaluating PCSK9 Binding antiBody Influence oN coGnitive HeAlth in High cardiovascUlar Risk Subjects
Acronym: EBBINGHAUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 20130385; 2014-001976-75 (EudraCT Number)
Record Dates: First submitted 2014-07-31; First posted 2014-08-04 (Estimated); Results first posted 2018-01-16 (Actual); Last update posted 2018-01-16 (Actual); Status verified 2017-12

CONDITIONS: Dyslipidemia
Keywords: High cholesterol; Treatment for high cholesterol; Lowering cholesterol; Lowering high cholesterol; Hypercholesterolemia
MeSH Terms: conditions — Dyslipidemias; Hypercholesterolemia | interventions — evolocumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Participants received placebo subcutaneous injections either once every 2 weeks (Q2W) or once a month (QM) according to their own preference. Participants continued with their background statin therapy during the course of the study.
  Interventions: Drug: Placebo; Drug: Background Statin Therapy
- Evolocumab (Experimental): Participants received evolocumab 140 mg Q2W or 420 mg QM subcutaneous injections according to their own preference. Participants continued with their background statin therapy during the course of the study.
  Interventions: Biological: Evolocumab; Drug: Background Statin Therapy

INTERVENTIONS:
Biological: Evolocumab — Administered subcutaneously using a spring-based prefilled 1.0 mL autoinjector/pen.
  Other Names: AMG 145; Repatha
  Arms: Evolocumab
Drug: Placebo — Administered subcutaneously using a spring-based prefilled 1.0 mL autoinjector/pen.
  Arms: Placebo
Drug: Background Statin Therapy — Participants were required to be on a stable, high- to moderate-intensity statin background therapy consisting of an effective statin dose, ie, at least atorvastatin 20 mg daily or equivalent, and where locally approved, highly effective statin therapy (defined as at least atorvastatin 40 mg daily or equivalent) was recommended.

SUMMARY:
This study evaluated change over time in neurocognitive testing in patients receiving statin therapy in combination with evolocumab (AMG 145), compared with patients receiving statin therapy in combination with placebo.

DETAILED DESCRIPTION:
Participants who were enrolled in study 20110118 (FOURIER; NCT01764633) at select sites in select countries (selected based on study start-up timelines) were invited to participate in this cognitive function study, 20130385. There was no separate randomization for Study 20130385; data were analyzed according to Study 20110118 randomized treatment arm.

ELIGIBILITY:
Inclusion Criteria:

* Randomized into Study 20110118 (FOURIER; NCT01764633)

Exclusion Criteria:

* Current or known past diagnosis of dementia or mild cognitive impairment (MCI)

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1974 (Actual)
Dates: Start 2014-09-10 (Actual); Primary Completion 2016-11-11 (Actual); Study Completion 2016-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (365):
- United States (126):
  - Research Site, Birmingham, Alabama
  - Research Site, Huntsville, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Glendale, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Alhambra, California
  - Research Site, Banning, California
  - Research Site, Harbor City, California
  - Research Site, Laguna Hills, California
  - Research Site, Long Beach, California
  - Research Site, Oceanside, California
  - Research Site, Oxnard, California
  - Research Site, Palm Springs, California
  - Research Site, Roseville, California
  - Research Site, Sacramento, California
  - Research Site, San Pedro, California
  - Research Site, Tarzana, California
  - Research Site, Thousand Oaks, California
  - Research Site, Aurora, Colorado
  - Research Site, Colorado Springs, Colorado
  - Research Site, Denver, Colorado
  - Research Site, Bridgeport, Connecticut
  - Research Site, Boynton Beach, Florida
  - Research Site, Crystal River, Florida
  - Research Site, Daytona Beach, Florida
  - Research Site, Deerfield Beach, Florida
  - Research Site, Fleming Island, Florida
  - Research Site, Hollywood, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Palm Harbor, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Ponte Vedra, Florida
  - Research Site, Sarasota, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Tampa, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Augusta, Georgia
  - Research Site, Gainesville, Georgia
  - Research Site, Savannah, Georgia
  - Research Site, Suwanee, Georgia
  - Research Site, Coeur d'Alene, Idaho
  - Research Site, Addison, Illinois
  - Research Site, Belleville, Illinois
  - Research Site, Chicago, Illinois
  - Research Site, Jerseyville, Illinois
  - Research Site, Hammond, Indiana
  - Research Site, Waterloo, Iowa
  - Research Site, Hutchinson, Kansas
  - Research Site, Lexington, Kentucky
  - Research Site, Owensboro, Kentucky
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Hammond, Louisiana
  - Research Site, Lafayette, Louisiana
  - Research Site, Metairie, Louisiana
  - Research Site, Monroe, Louisiana
  - Research Site, Slidell, Louisiana
  - Research Site, Biddeford, Maine
  - Research Site, Salisbury, Maryland
  - Research Site, Towson, Maryland
  - Research Site, Haverhill, Massachusetts
  - Research Site, Newton, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Grandville, Michigan
  - Research Site, Lansing, Michigan
  - Research Site, Muskegon, Michigan
  - Research Site, Saint Paul, Minnesota
  - Research Site, Jefferson City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Great Falls, Montana
  - Research Site, Kalispell, Montana
  - Research Site, Voorhees Township, New Jersey
  - Research Site, Westwood, New Jersey
  - Research Site, Brooklyn, New York
  - Research Site, Buffalo, New York
  - Research Site, Cortlandt Manor, New York
  - Research Site, New Hyde Park, New York
  - Research Site, New Windsor, New York
  - Research Site, Rochester, New York
  - Research Site, Troy, New York
  - Research Site, West Seneca, New York
  - Research Site, Williamsville, New York
  - Research Site, Calabash, North Carolina
  - Research Site, Hickory, North Carolina
  - Research Site, Mooresville, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Tabor City, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Grand Forks, North Dakota
  - Research Site, Canton, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Springfield, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Pryor, Oklahoma
  - Research Site, Bend, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Camp Hill, Pennsylvania
  - Research Site, Chambersburg, Pennsylvania
  - Research Site, Feasterville, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Pawtucket, Rhode Island
  - Research Site, Fort Mill, South Carolina
  - Research Site, Moncks Corner, South Carolina
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, North Myrtle Beach, South Carolina
  - Research Site, Rapid City, South Dakota
  - Research Site, Jackson, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Tullahoma, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Plano, Texas
  - Research Site, Wichita Falls, Texas
  - Research Site, West Jordan, Utah
  - Research Site, Burke, Virginia
  - Research Site, Falls Church, Virginia
  - Research Site, Hopewell, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Suffolk, Virginia
  - Research Site, Seattle, Washington
  - Research Site, Green Bay, Wisconsin
- Australia (9):
  - Research Site, Woden, Australian Capital Territory
  - Research Site, Auchenflower, Queensland
  - Research Site, Adelaide, South Australia
  - Research Site, Ashford, South Australia
  - Research Site, Fullarton, South Australia
  - Research Site, Hobart, Tasmania
  - Research Site, Box Hill, Victoria
  - Research Site, Epping, Victoria
  - Research Site, Geelong, Victoria
- Belgium (7):
  - Research Site, Aalst
  - Research Site, Bonheiden
  - Research Site, Brussels
  - Research Site, Gozée
  - Research Site, Ieper
  - Research Site, La Louvière
  - Research Site, Liège
- Canada (11):
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, London, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, Peterborough, Ontario
  - Research Site, Sarnia, Ontario
  - Research Site, Chicoutimi, Quebec
  - Research Site, Gatineau, Quebec
  - Research Site, Pointe-Claire, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Saint-Jean-sur-Richelieu, Quebec
  - Research Site, Saint-Jérôme, Quebec
- Czechia (18):
  - Research Site, Beroun
  - Research Site, Bílovec
  - Research Site, Brandýs nad Labem
  - Research Site, Brno
  - Research Site, Chomutov
  - Research Site, Havlíčkův Brod
  - Research Site, Hodonín
  - Research Site, Klatovy IV
  - Research Site, Liberec
  - Research Site, Litomyšl
  - Research Site, Mohelnice
  - Research Site, Olomouc
  - Research Site, Ostrava - Vitkovice
  - Research Site, Pardubice
  - Research Site, Prague
  - Research Site, Praha 5 - Smichov
  - Research Site, Přerov
  - Research Site, Uherské Hradiště
- Denmark (7):
  - Research Site, Aalborg
  - Research Site, Ballerup Municipality
  - Research Site, Esbjerg
  - Research Site, Hvidovre
  - Research Site, København S
  - Research Site, Køge
  - Research Site, Vejle
- Estonia (2):
  - Research Site, Paide
  - Research Site, Tallinn
- Finland (7):
  - Research Site, Helsinki
  - Research Site, Jyväskylä
  - Research Site, Kuopio
  - Research Site, Oulu
  - Research Site, OYS
  - Research Site, Tampere
  - Research Site, Turku
- France (7):
  - Research Site, Besançon
  - Research Site, Le Coudray
  - Research Site, Montepellier Cedex
  - Research Site, Nantes
  - Research Site, Paris
  - Research Site, Pessac
  - Research Site, Toulouse
- Germany (12):
  - Research Site, Bad Krozingen
  - Research Site, Berlin
  - Research Site, Bochum
  - Research Site, Cologne
  - Research Site, Dresden
  - Research Site, Frankfurt am Main
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Leipzig
  - Research Site, Stuttgart
  - Research Site, Witten
  - Research Site, Wuppertal
- Greece (5):
  - Research Site, Alexandroupoli
  - Research Site, Athens
  - Research Site, Ioannina
  - Research Site, Larissa
  - Research Site, Piraeus
- Research Site, Hong Kong, Hong Kong
- Hungary (9):
  - Research Site, Berettyóújfalu
  - Research Site, Békéscsaba
  - Research Site, Budapest
  - Research Site, Nyíregyháza
  - Research Site, Pécs
  - Research Site, Szeged
  - Research Site, Szekszárd
  - Research Site, Szikszó
  - Research Site, Zalaegerszeg
- Research Site, Pavia, Italy
- Japan (22):
  - Research Site, Ichinomiya-shi, Aichi-ken
  - Research Site, Kasugai-shi, Aichi-ken
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Toyohashi, Aichi-ken
  - Research Site, Matsudo-shi, Chiba
  - Research Site, Saijo-shi, Ehime
  - Research Site, Chikushi-gun, Fukuoka
  - Research Site, Fukuoka, Fukuoka
  - Research Site, Itoshima-shi, Fukuoka
  - Research Site, Sapporo, Hokkaido
  - Research Site, Himeji-shi, Hyōgo
  - Research Site, Toride-shi, Ibaraki
  - Research Site, Tsukuba, Ibaraki
  - Research Site, Kyoto, Kyoto
  - Research Site, Okinawa-shi, Okinawa
  - Research Site, Shimajiri-gun, Okinawa
  - Research Site, Urasoe-shi, Okinawa
  - Research Site, Osaka, Osaka
  - Research Site, Saga, Saga-ken
  - Research Site, Kawaguchi-shi, Saitama
  - Research Site, Komatsushima-shi, Tokushima
  - Research Site, Chuo-ku, Tokyo
- Latvia (5):
  - Research Site, Daugavpils
  - Research Site, Kuldīga
  - Research Site, Liepāja
  - Research Site, Ogre
  - Research Site, Riga
- Research Site, Vilnius, Lithuania
- Malaysia (2):
  - Research Site, Kuala Lumpur, Kuala Lumpur
  - Research Site, Kuala Lumpur
- Netherlands (5):
  - Research Site, Arnhem
  - Research Site, Ede
  - Research Site, Eindhoven
  - Research Site, Hoorn
  - Research Site, Uden
- New Zealand (2):
  - Research Site, Christchurch
  - Research Site, Tauranga
- Norway (7):
  - Research Site, Ålesund
  - Research Site, Hamar
  - Research Site, Lierskogen
  - Research Site, Oslo
  - Research Site, Skedsmokorset
  - Research Site, Skien
  - Research Site, Stavanger
- Poland (19):
  - Research Site, Gdansk
  - Research Site, Gdynia
  - Research Site, Katowice
  - Research Site, Kielce
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Olsztyn
  - Research Site, Poznan
  - Research Site, Puławy
  - Research Site, Ruda Śląska
  - Research Site, Staszów
  - Research Site, Świdnik
  - Research Site, Tarnów
  - Research Site, Torun
  - Research Site, Warsaw
  - Research Site, Wroclaw
  - Research Site, Włocławek
  - Research Site, Zamość
- Portugal (4):
  - Research Site, Almada
  - Research Site, Carnaxide
  - Research Site, Coimbra
  - Research Site, Covilha
- Russia (13):
  - Research Site, Ivanovo
  - Research Site, Izhevsk
  - Research Site, Kemerovo
  - Research Site, Kirov
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Omsk
  - Research Site, Pushkin
  - Research Site, Saint Petersburg
  - Research Site, Saratov
  - Research Site, Tomsk
  - Research Site, Yekaterinburg
- Slovakia (12):
  - Research Site, Bardejov
  - Research Site, Brezno
  - Research Site, Košice
  - Research Site, Lučenec
  - Research Site, Moldava nad Bodvou
  - Research Site, Nové Zámky
  - Research Site, Rimavská Sobota
  - Research Site, Rožňava
  - Research Site, Snina
  - Research Site, Svidník
  - Research Site, Trenčín
  - Research Site, Trnava
- South Africa (10):
  - Research Site, Centurion, Gauteng
  - Research Site, Johannesburg, Gauteng
  - Research Site, Pretoria, Gauteng
  - Research Site, Pretoria West, Gauteng
  - Research Site, Paarl, Western Cape
  - Research Site, Parow, Western Cape
  - Research Site, Somerset West, Western Cape
  - Research Site, Worcester, Western Cape
  - Research Site, Cape Town
  - Research Site, Kempton Park
- Spain (7):
  - Research Site, Zaragoza, Aragon
  - Research Site, Galdakao, Basque Country
  - Research Site, L'Hospitalet de Llobregat, Catalonia
  - Research Site, Santiago de Compostela, Galicia
  - Research Site, Vigo, Galicia
  - Research Site, Valencia, Valencia
  - Research Site, Madrid
- Sweden (6):
  - Research Site, Helsingborg
  - Research Site, Linköping
  - Research Site, Lund
  - Research Site, Stockholm
  - Research Site, Uddevalla
  - Research Site, Västerås
- Turkey (Türkiye) (6):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Gaziantep
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Kocaeli
- United Kingdom (22):
  - Research Site, Belfast
  - Research Site, Birmingham
  - Research Site, Bournemouth
  - Research Site, Cardiff
  - Research Site, Chesterfield
  - Research Site, Chippenham
  - Research Site, Chorley
  - Research Site, Doncaster
  - Research Site, Glasgow
  - Research Site, Hexham
  - Research Site, Leicester
  - Research Site, Liverpool
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Newport
  - Research Site, Nuneaton
  - Research Site, Reading
  - Research Site, Sandbach
  - Research Site, Sheffield
  - Research Site, West Bromwich
  - Research Site, Whitby
  - Research Site, Worcester

REFERENCES:
- [Background] Giugliano RP, Mach F, Zavitz K, Kurtz C, Schneider J, Wang H, Keech A, Pedersen TR, Sabatine MS, Sever PS, Honarpour N, Wasserman SM, Ott BR; EBBINGHAUS Investigators. Design and rationale of the EBBINGHAUS trial: A phase 3, double-blind, placebo-controlled, multicenter study to assess the effect of evolocumab on cognitive function in patients with clinically evident cardiovascular disease and receiving statin background lipid-lowering therapy-A cognitive study of patients enrolled in the FOURIER trial. Clin Cardiol. 2017 Feb;40(2):59-65. doi: 10.1002/clc.22678. Epub 2017 Feb 16. PMID 28207168
- [Background] Giugliano RP, Mach F, Zavitz K, Kurtz C, Im K, Kanevsky E, Schneider J, Wang H, Keech A, Pedersen TR, Sabatine MS, Sever PS, Robinson JG, Honarpour N, Wasserman SM, Ott BR; EBBINGHAUS Investigators. Cognitive Function in a Randomized Trial of Evolocumab. N Engl J Med. 2017 Aug 17;377(7):633-643. doi: 10.1056/NEJMoa1701131. PMID 28813214
- [Derived] Schmidt AF, Carter JL, Pearce LS, Wilkins JT, Overington JP, Hingorani AD, Casas JP. PCSK9 monoclonal antibodies for the primary and secondary prevention of cardiovascular disease. Cochrane Database Syst Rev. 2020 Oct 20;10(10):CD011748. doi: 10.1002/14651858.CD011748.pub3. PMID 33078867
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled in Study 20110118 (FOURIER; NCT01764633) at select sites in select countries (based on study start-up timelines) were invited to participate in this cognitive function study.
  Participants were enrolled at 340 centers in 29 countries in Europe, North America, and Asia Pacific from September 2014 to July 2015.
Pre-assignment Details: There was no separate randomization in this study; each participant received their assigned treatment per Protocol 20110118. Data were analyzed according to Study 20110118 randomized treatment arm.
Period: Overall Study
Arm/Group | Placebo | Evolocumab
Started | 990 | 984
Received Treatment | 990 | 983
Completed | 968 | 953
Not Completed | 22 | 31
Not completed — Withdrawal by Subject | 21 | 31
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Demographic data are provided for all enrolled participants. Baseline Cambridge Neuropsychological Test Automated Battery (CANTAB®) data are provided for all dosed participants enrolled in the study with a baseline cognitive function assessment prior to or on the first dose date of study drug and ≥ 1 post-baseline cognitive measure.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Evolocumab | Total
Number analyzed (Participants) | 990 | 984 | 1974
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (8.7) | 62.9 (8.7) | 62.8 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 274 | 269 | 543
  Male | 716 | 715 | 1431
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 9 | 23
  Not Hispanic or Latino | 976 | 975 | 1951
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 28 | 31 | 59
  Black or African American | 32 | 28 | 60
  Native Hawaiian or Other Pacific Islander | 0 | 3 | 3
  White | 910 | 908 | 1818
  Multiple | 1 | 1 | 2
  Other | 17 | 12 | 29
Spatial Working Memory (SWM) Strategy Index of Executive Function Raw Score [Mean (Standard Deviation); unit: units on a scale] — CANTAB is a series of computerized tests to assess cognitive function. The SWM test assesses the cognitive domain of executive function (high-level thinking and decision making). Patients search for colored tokens hidden inside boxes on the screen. Tokens were never hidden inside the same box twice, so patients must not return to a box where a token was already found. The SWM strategy index of executive function represents the number of times a patient began a search with a different box. A high score represents an inefficient use of strategy and planning. The raw score ranges from 4 to 28. Population: All enrolled and dosed participants who completed a baseline cognitive functional assessment prior to or on the first date of administration of study drug and who have at least one post-baseline cognitive measure.
  units on a scale
    number analyzed (Participants) | 618 | 586 | 1204
    (all) | 17.8 (3.4) | 17.8 (3.5) | 17.8 (3.4)
Spatial Working Memory (SWM) Strategy Index of Executive Function Z Score [Mean (Standard Deviation); unit: Z score] — The CANTAB SWM test assesses the cognitive domain of executive function (high-level thinking and decision making). Patients search for colored tokens hidden inside boxes on the screen. Tokens were never hidden inside the same box twice, so patients must not return to a box where a token was already found. The SWM strategy index of executive function represents the number of times a patient began a search with a different box. The Z score represents the standardized measure of how far an individual deviates from the study cohort average at baseline. A higher Z score reflects better performance. Population: All enrolled and dosed participants who completed a baseline cognitive functional assessment prior to or on the first date of administration of study drug and who have at least one post-baseline cognitive measure.
  Z score
    number analyzed (Participants) | 618 | 586 | 1204
    (all) | -0.0106 (0.9910) | 0.0166 (1.0066) | 0.0026 (0.9983)
Spatial Working Memory Between Errors Raw Score [Mean (Standard Deviation); unit: units on a scale] — The CANTAB Spatial Working Memory (SWM) between-errors score test assesses the cognitive domain of working memory (holding material in mind while that material is being actively processed). Patients search for colored tokens hidden inside boxes on the screen. Tokens were never hidden inside the same box twice, so patients must not return to a box where a token was already found. The SWM between-errors score is the number of times that a patient revisited a box in which a token had previously been found. A lower score indicates better performance. The raw score ranges from 0 to 279. Population: All enrolled and dosed participants who completed a baseline cognitive functional assessment prior to or on the first date of administration of study drug and who have at least one post-baseline cognitive measure.
  units on a scale
    number analyzed (Participants) | 618 | 586 | 1204
    (all) | 21.0 (10.6) | 20.9 (10.2) | 21.0 (10.4)
Spatial Working Memory Between Errors Z Score [Mean (Standard Deviation); unit: Z score] — The CANTAB Spatial Working Memory (SWM) between-errors score test assesses the cognitive domain of working memory (holding material in mind while that material is being actively processed). Patients search for colored tokens hidden inside boxes on the screen. Tokens were never hidden inside the same box twice, so patients must not return to a box where a token was already found The SWM between-errors score is the number of times a patient revisited a box in which a token had already been found. A higher Z score reflects better performance. Population: All enrolled and dosed participants who completed a baseline cognitive functional assessment prior to or on the first date of administration of study drug and who have at least one post-baseline cognitive measure.
  Z score
    number analyzed (Participants) | 618 | 586 | 1204
    (all) | -0.0130 (1.0075) | 0.0024 (0.9675) | -0.0055 (0.9879)
Paired Associates Learning (PAL) Total Errors Adjusted Raw Score [Mean (Standard Deviation); unit: units on a scale] — The CANTAB PAL test assesses memory function (storing/retrieving information by associating an event with a time and place). Boxes on the screen open in turn to reveal a number of patterns. After all the boxes were opened, each pattern was shown in a randomized order and the patient asked to touch the box where they think the pattern was hidden. The PAL total errors adjusted score is the number of errors made plus an adjustment for the estimated number of errors the patient would have made on any stages not reached. A lower score indicates better performance. The raw score ranges from 0 to 70. Population: All enrolled and dosed participants who completed a baseline cognitive functional assessment prior to or on the first date of administration of study drug and who have at least one post-baseline cognitive measure.
  units on a scale
    number analyzed (Participants) | 618 | 586 | 1204
    (all) | 25.2 (18.4) | 26.5 (19.3) | 25.8 (18.9)
Paired Associates Learning Total Errors Adjusted Z Score [Mean (Standard Deviation); unit: Z score] — The CANTAB PAL test assesses memory function (storing/retrieving information by associating an event with a time and place). Boxes on the screen open in turn to reveal a number of patterns. After all the boxes have been opened, each pattern was shown in a randomized order and the patient asked to touch the box where they think each pattern was hidden. The PAL total errors adjusted is the number of errors committed plus an adjustment for the estimated number of errors the patient would have made on any stages not reached. Higher Z scores indicate better performance. Population: All enrolled and dosed participants who completed a baseline cognitive functional assessment prior to or on the first date of administration of study drug and who have at least one post-baseline cognitive measure.
  Z score
    number analyzed (Participants) | 618 | 586 | 1204
    (all) | 0.0442 (0.9834) | -0.0272 (1.0294) | 0.0095 (1.0063)
Reaction Time Median 5-Choice Reaction Time Raw Score [Mean (Standard Deviation); unit: msec] — The CANTAB Reaction Time (RTI) test assessed psychomotor speed (detecting and responding to a stimulus). Participants held down a button until a spot appeared in 1 of 5 circles on the screen. As soon as possible after the spot flashed up, the patient lifted their finger from the button and touched the circle in which the spot appeared. The RTI median 5-choice reaction time was the median duration between the onset of the stimulus and the release of the button. A lower score indicates better performance. The raw score ranges from 100 to 5100 msec. Population: All enrolled and dosed participants who completed a baseline cognitive functional assessment prior to or on the first date of administration of study drug and who have at least one post-baseline cognitive measure.
  msec
    number analyzed (Participants) | 614 | 585 | 1199
    (all) | 355.10 (77.60) | 356.74 (65.01) | 355.90 (71.71)
Reaction Time Median 5-Choice Reaction Time Z Score [Mean (Standard Deviation); unit: Z-score] — The CANTAB Reaction Time (RTI) test assessed psychomotor speed (detecting and responding to a stimulus). Participants held down a button until a spot appeared in 1 of 5 circles on the screen. As soon as possible after the spot flashed up, the patient moved their finger from the button to the circle in which the spot appeared. The RTI median 5-choice reaction time is the median duration between the onset of the stimulus and the release of the button. A higher Z score reflects better performance. Population: All enrolled and dosed participants who completed a baseline cognitive functional assessment prior to or on the first date of administration of study drug and who have at least one post-baseline cognitive measure.
  Z-score
    number analyzed (Participants) | 614 | 585 | 1199
    (all) | -0.0271 (1.0829) | -0.0500 (0.9072) | -0.0383 (1.0007)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Spatial Working Memory Strategy Index of Executive Function (6-8 Boxes) Z Score
Description: Assessments were performed with the Cambridge Neuropsychological Test Automated Battery (CANTAB), a language-independent battery of computerized tests that is used to assess cognitive function.
  The Spatial Working Memory (SWM) test assesses the cognitive domain of executive function (high-level thinking and decision making). Patients search for colored tokens hidden inside boxes on the screen by touching them. The critical instruction is that once a token has been found inside a box, there will never be a token hidden inside that box again, so patients must not return to a box where a token has been found.
  The SWM strategy index of executive function represented the number of times a subject began a search with a different box. The Z score represents the standardized measure of how far an individual subject deviates from the study cohort average at baseline. A higher Z score reflects better performance. The mean change from baseline averaged across all the visits is reported.
Time Frame: Assessments were conducted at Baseline and at weeks 24, 48, 96, 144 and end of study visit (median time on study was 19.4 months).
Population: All enrolled and dosed participants who completed a baseline cognitive functional assessment prior to or on the first date of administration of study drug and who have at least one post-baseline cognitive measure.
  Cognitive function assessments after an on-study stroke event were excluded from the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Z score
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 616 | 586
Z score | 0.1206 [0.0535 to 0.1877] | 0.1134 [0.0449 to 0.1820]
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; A repeated measures mixed-effect linear model was used to estimate treatment difference (placebo - evolocumab) in change from baseline and associated 95% confidence intervals (CI). The model included stratification factors for Study 20110118 (final screening low-density lipoprotein cholesterol [LDL-C] and geographical region), age, education level, baseline SWM strategy index Z score, treatment group, visit, and treatment by visit interaction; Test type: Non-Inferiority — The non-inferiority margin was 0.19, calculated as 20% of the observed common standard deviation, which was estimated from observations in the placebo group by a repeated measured mixed-effect linear model with visit as a covariate. If the upper bound of the 95% CI for the difference between the placebo and evolocumab group in mean change from baseline for Z score averaged across the visits was less than the non-inferiority margin non-inferiority criteria were met; Treatment Difference = 0.0072, 95% CI 2-sided [-0.0664 to 0.0808], Standard Error of Mean 0.0375

2. Secondary Outcome: Mean Change From Baseline in Spatial Working Memory (SWM) Between-errors Z Score
Description: Assessments were performed with the CANTAB, a language-independent battery of computerized tests that is used to assess cognitive function. The Spatial Working Memory (SWM) between-errors test assesses the cognitive domain of working memory (holding material in mind while that material is being actively processed). Patients search for colored tokens hidden inside boxes on the screen by touching them. The critical instruction is that once a token has been found inside a box, there will never be a token hidden inside that box again, so patients must not return to a box where a token has been found.
  The SWM between-errors score is the number of times that a patient revisited a box in which a token had previously been found. The Z score represents the standardized measure of how far an individual participant deviates from the study cohort average at baseline. A higher Z score reflects better performance. The mean change from baseline averaged across all the visits is reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Z score
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 616 | 586
Z score | 0.1024 [0.0373 to 0.1675] | 0.0691 [0.0026 to 0.1355]
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; A repeated measures mixed-effect linear model was used to estimate treatment difference (placebo - evolocumab) in change from baseline and associated 95% confidence intervals (CI). The model included stratification factors for Study 20110118 (final screening LDL-C and geographical region), age, education level, baseline SWM between-errors Z score, treatment group, visit, and treatment by visit interaction; Test type: Other; Treatment Difference = 0.0333, 95% CI 2-sided [-0.0378 to 0.1045], Standard Error of Mean 0.0363

3. Secondary Outcome: Mean Change From Baseline in Paired Associated Learning (PAL) Total Errors Adjusted Z Score
Description: The CANTAB PAL test assesses visuospatial episodic memory (storing/retrieving information by associating an event with a time and place). Boxes on the screen opened up one at a time to reveal a number of patterns. Participants were asked to remember the location of each pattern. After all the boxes had been opened, each pattern was then shown in the center of the screen in a randomized order, and the patient should touch the box where they think each pattern was hidden. The PAL total errors adjusted comprised the number of errors committed by a patient plus an adjustment for the estimated number of errors the patient would have made on any stages that were not reached.
  Z score represents the standardized measure of how far an individual patient deviates from the study cohort average at baseline. A higher Z score indicated better performance. The mean change from baseline averaged across all the visits is reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Z score
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 615 | 585
Z score | 0.1098 [0.0511 to 0.1686] | 0.0873 [0.0273 to 0.1472]
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; A repeated measures mixed-effect linear model was used to estimate treatment difference (placebo - evolocumab) in change from baseline and associated 95% confidence intervals (CI). The model included stratification factors for Study 20110118 (final screening LDL-C and geographical region), age, education level, baseline PAL total errors adjusted Z score, treatment group, visit, and treatment by visit interaction; Test type: Other; Treatment Difference = 0.0226, 95% CI 2-sided [-0.0422 to 0.0873], Standard Error of Mean 0.0330

4. Secondary Outcome: Mean Change From Baseline in Reaction Time (RTI) Median 5-choice Reaction Time Z Score
Description: Assessments were performed with the CANTAB, a language-independent battery of computerized tests that is used to assess cognitive function. The Reaction Time (RTI) test assessed the cognitive domain of psychomotor speed (detecting and responding to a stimulus). Participants held down a button until a spot appeared in 1 of 5 circles on the screen. As soon as possible after the spot flashed up, the patient lifted their finger from the button and touched the circle in which the spot appeared. The RTI median 5-choice reaction time was the median duration between the onset of the stimulus and the release of the button. Z score represents the standardized measure of how far an individual participant deviates from the study cohort average at baseline. A higher Z score reflects better performance. The mean change from baseline averaged across all the visits is reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Z score
Arm/Group | Placebo | Evolocumab
Number analyzed (Participants) | 611 | 584
Z score | 0.0153 [-0.0529 to 0.0834] | -0.0575 [-0.1270 to 0.0121]
Statistical Analysis 1: Comparison: Placebo vs Evolocumab; A repeated measures mixed-effect linear model was used to estimate treatment difference ( placebo - evolocumab) in change from baseline and associated 95% confidence intervals (CI). The model included stratification factors for Study 20110118 (final screening LDL-C and geographical region), age, education level, baseline RTI median 5-choice reaction time Z score, treatment group, visit, and treatment by visit interaction; Test type: Other; Treatment Difference = 0.0727, 95% CI 2-sided [-0.0022 to 0.1477], Standard Error of Mean 0.0382

ADVERSE EVENTS:
Time Frame: From the first dose of study drug to the end of study. The median duration of follow-up was 19.4 months.
Description: Although there was no separate safety data collection, recording, or reporting planned in this study, an ad-hoc analysis of safety data collected in Study 20110118 was conducted for participants in Study 20130385 and is reported here.
  Deaths by any cause were collected as adjudicated efficacy endpoints in Study 20110118 and were reported as a secondary endpoint in Study 20110118.
  Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the 5% frequency threshold.
Arm/Group | Placebo | Evolocumab
Serious Adverse Events (participants affected / at risk) | 204/990 | 212/983
Other Adverse Events (participants affected / at risk) | 257/990 | 272/983
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=990) | Evolocumab (N=983)
Anaemia (Blood and lymphatic system disorders) | 6 | 2
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 1
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 1
Spleen disorder (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 16 | 15
Angina unstable (Cardiac disorders) | 15 | 11
Arrhythmia (Cardiac disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 7 | 13
Atrial flutter (Cardiac disorders) | 1 | 1
Atrioventricular block (Cardiac disorders) | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 3 | 0
Bundle branch block left (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 4 | 1
Cardiac failure acute (Cardiac disorders) | 1 | 1
Cardiac failure chronic (Cardiac disorders) | 4 | 2
Cardiac failure congestive (Cardiac disorders) | 5 | 4
Cardiac tamponade (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1
Congestive cardiomyopathy (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 3 | 2
Dressler's syndrome (Cardiac disorders) | 1 | 0
Heart alternation (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Left ventricular failure (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 3
Mitral valve stenosis (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Myocarditis (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 1
Sinus arrest (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1
Sinus node dysfunction (Cardiac disorders) | 1 | 1
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 3 | 1
Intracranial lipoma (Congenital, familial and genetic disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 1
Cataract (Eye disorders) | 2 | 0
Iridocyclitis (Eye disorders) | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0
Strabismus (Eye disorders) | 1 | 0
Uveitis (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 2
Abdominal pain lower (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Coeliac artery stenosis (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Diverticulum (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 1
Gastric disorder (Gastrointestinal disorders) | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 1
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 2 | 2
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 3
Large intestine polyp (Gastrointestinal disorders) | 1 | 0
Mesenteric artery stenosis (Gastrointestinal disorders) | 0 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 1
Pancreatic cyst (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Peptic ulcer (Gastrointestinal disorders) | 1 | 0
Reflux gastritis (Gastrointestinal disorders) | 0 | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 4 | 2
Non-cardiac chest pain (General disorders) | 12 | 6
Oedema peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Soft tissue inflammation (General disorders) | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholangitis acute (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 1 | 1
Cholelithiasis obstructive (Hepatobiliary disorders) | 0 | 1
Liver disorder (Hepatobiliary disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Appendiceal abscess (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 2 | 0
Burkholderia cepacia complex infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 1
Clostridium difficile infection (Infections and infestations) | 1 | 1
Cystitis (Infections and infestations) | 0 | 1
Device related sepsis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Escherichia sepsis (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 1
Hepatitis C (Infections and infestations) | 0 | 1
Hepatitis E (Infections and infestations) | 1 | 1
Infectious pleural effusion (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 0
Lung infection (Infections and infestations) | 1 | 0
Mastoiditis (Infections and infestations) | 1 | 0
Orchitis (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 2 | 3
Peritonitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 7 | 10
Pneumonia bacterial (Infections and infestations) | 1 | 2
Post procedural sepsis (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 4 | 0
Septic shock (Infections and infestations) | 1 | 0
Streptococcal sepsis (Infections and infestations) | 1 | 0
Upper respiratory tract infection bacterial (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 2
Urinary tract infection bacterial (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 2 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 0
Arterial bypass occlusion (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 2
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 | 1
Dislocation of sternum (Injury, poisoning and procedural complications) | 0 | 1
Eye injury (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 2
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1
Peripheral arterial reocclusion (Injury, poisoning and procedural complications) | 0 | 1
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 1 | 1
Pneumoconiosis (Injury, poisoning and procedural complications) | 0 | 1
Pneumonitis chemical (Injury, poisoning and procedural complications) | 0 | 1
Post concussion syndrome (Injury, poisoning and procedural complications) | 0 | 1
Post procedural constipation (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Post procedural swelling (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal column injury (Injury, poisoning and procedural complications) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 0
Arteriogram coronary (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 3 | 0
Blood potassium increased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 2
Liver function test abnormal (Investigations) | 0 | 1
Myocardial necrosis marker increased (Investigations) | 1 | 0
Thyroid function test abnormal (Investigations) | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 2
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Myalgia intercostal (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder transitional cell carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Laryngeal cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lip and/or oral cavity cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1
Lung squamous cell carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Arachnoid cyst (Nervous system disorders) | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 1
Carotid artery disease (Nervous system disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 5 | 6
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Cervical myelopathy (Nervous system disorders) | 0 | 1
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 2
Facial paralysis (Nervous system disorders) | 1 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1
Guillain-Barre syndrome (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 3 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1
Meralgia paraesthetica (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Paraparesis (Nervous system disorders) | 0 | 1
Parkinsonism (Nervous system disorders) | 1 | 0
Radiculopathy (Nervous system disorders) | 1 | 1
Sciatica (Nervous system disorders) | 2 | 0
Seizure (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 4 | 3
Transient ischaemic attack (Nervous system disorders) | 1 | 2
Device malfunction (Product Issues) | 2 | 0
Device occlusion (Product Issues) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Major depression (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 6 | 2
Calculus urethral (Renal and urinary disorders) | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 2 | 0
End stage renal disease (Renal and urinary disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 1 | 2
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 2 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 1
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma-chronic obstructive pulmonary disease overlap syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 2
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 2 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 2
Fracture treatment (Surgical and medical procedures) | 1 | 0
Gastric banding reversal (Surgical and medical procedures) | 1 | 0
Accelerated hypertension (Vascular disorders) | 0 | 1
Aortic aneurysm (Vascular disorders) | 4 | 1
Aortic aneurysm rupture (Vascular disorders) | 1 | 0
Aortic stenosis (Vascular disorders) | 1 | 0
Arterial occlusive disease (Vascular disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 2
Hypertension (Vascular disorders) | 5 | 7
Hypertensive crisis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 3
Iliac artery occlusion (Vascular disorders) | 1 | 0
Intermittent claudication (Vascular disorders) | 2 | 2
Leriche syndrome (Vascular disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 5 | 10
Peripheral artery occlusion (Vascular disorders) | 1 | 0
Peripheral artery stenosis (Vascular disorders) | 4 | 2
Peripheral artery thrombosis (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 4 | 6
Peripheral vascular disorder (Vascular disorders) | 1 | 1
Subclavian artery stenosis (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 2 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=990) | Evolocumab (N=983)
Nasopharyngitis (Infections and infestations) | 74 | 101
Upper respiratory tract infection (Infections and infestations) | 63 | 53
Diabetes mellitus (Metabolism and nutrition disorders) | 59 | 45
Back pain (Musculoskeletal and connective tissue disorders) | 36 | 58
Hypertension (Vascular disorders) | 66 | 61

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.